CLINICAL TRIAL: NCT01380704
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Safety and Pharmacodynamic Effects of ABT-436 in Major Depressive Disorder Subjects
Brief Title: Safety and Pharmacodynamic Study of ABT-436 in Major Depressive Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M12-674
Record Dates: First submitted 2011-06-01; First posted 2011-06-27 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2011-11

CONDITIONS: Major Depressive Disorder
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: ABT-436
- Placebo (Placebo Comparator)
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: ABT-436 — QD Days 1-7
  Arms: Active
Drug: Matching Placebo — QD Days 1-7
  Arms: Placebo

SUMMARY:
This is a multiple-dose study to assess the safety and pharmacology of ABT-436 in physically healthy subjects with mild to moderate depressive symptoms who are not taking any antidepressant medication. Efficacy for treatment of depressive symptoms is not a goal of this study.

DETAILED DESCRIPTION:
This is a multiple-dose study to assess the safety and pharmacology of ABT-436 in physically healthy subjects with mild to moderate depressive symptoms who are not taking any antidepressant medication. Efficacy for treatment of depressive symptoms is not a goal of this study. Fifty subjects will receive study drug for seven days. Thirty subjects will receive ABT-436 and twenty subjects will receive placebo. Blood, urine and saliva samples will be obtained, both before and during study drug administration, to measure ABT-436 pharmacology. Safety will be assessed throughout the study, including at two follow-up visits after completion of study drug administration.

ELIGIBILITY:
Inclusion Criteria

1. Age between 18 to 55 years, inclusive. 2. Body Mass Index is 20 to 35 kg/m2, inclusive. 3. A primary Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition, Text Revision (DSM-IV-TR) diagnosis of major depressive disorder.

4. Mild-to-moderate depressive symptoms at Screening. 5. A condition of general good physical health. Exclusion Criteria

1. Pregnant or breast-feeding female.
2. Use of any medication within 4 weeks prior to Day -2, unless the dose has been stable for 4 weeks, no dose change is anticipated during the study, and the medication is specifically allowed for this study, OR prior as needed (PRN) use of the medication is specifically allowed for this study.
3. Use of fluoxetine or aripiprazole within 8 weeks prior to Day -2.
4. Positive screen for drugs of abuse/alcohol, recent history of drug/alcohol abuse or smoking.
5. A current or past history of major depressive disorder with psychotic features, bipolar disorder, schizophrenia or other psychotic disorder, mental retardation, or mental disorder due to a general medical condition.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Pharmacology assays | Days -2, -1, 6, 7
  Hormones in blood, urine and saliva samples
ABT-436 drug levels | Days 6, 7
  ABT-436 drug levels in plasma
Vital signs | Days -2 through 8, 14, 30
  Blood pressure, pulse
Clinical safety labs | Days -2, 2, 5, 8
  Hematology, chemistry, urinalysis

SECONDARY OUTCOMES:
Psychiatric symptom scales | Days -2, 7
  Hamilton depression scale, Mood and anxiety symptom questionnaire, Perceived stress scale

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Tracy, MD, Study Director — Abbott

REFERENCES:
- [Result] Katz DA, Locke C, Greco N, Liu W, Tracy KA. Hypothalamic-pituitary-adrenal axis and depression symptom effects of an arginine vasopressin type 1B receptor antagonist in a one-week randomized Phase 1b trial. Brain Behav. 2017 Feb 9;7(3):e00628. doi: 10.1002/brb3.628. eCollection 2017 Mar. PMID 28293470